CLINICAL TRIAL: NCT04463849
Title: Effects of SARS-CoV-2 Infection on Beta-cell Function in Euglycemic Patients
Brief Title: Effects of COVID-19 Infection on Beta-cell Function in Euglycemic Patients
Acronym: COBETOX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Milan (Other)
Collaborators: Luigi Sacco University Hospital (Other)
Responsible Party: Principal Investigator, Paolo Fiorina, MD, Clinical Professor, University of Milan
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 6/2020
Record Dates: First submitted 2020-07-02; First posted 2020-07-09 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: COVID19; BETA-CELL FUNCTION
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- COVID-19 positive patients (Experimental): Patients will be enrolled in hospital for confirmed COVID-19 infection (with reverse transcriptase-polymerase chain reaction on the airway swab) but with normal basal glucose and no previous history of diabetes or impaired fasting glucose or impaired tolerance glucose. Patients will be placed with a professional retrospective glucose monitoring device and will be tested for stimulation with arginine infusion. The device will be placed on the day of the test and will be removed after seven days of recording the glycemic data. During the entire recording period, parameters such as mean glucose, estimated glycosylated hemoglobin, peak glucose and nadir, blood sugar levels above the limit of 140 mg / dL, average glucose values at 60 and 120 minutes after meals, standard deviation and variability coefficient.
  Interventions: Diagnostic Test: Stimulation test with arginine infusion in order to verify the possible existence of damage to the beta cell function induced by COVID-19 infection
- Healthy volunteers (Other): Healthy volunteers, not affected by COVID-19 and with no previous history of diabetes or impaired fasting glucose or impaired glucose tolerance will be enrolled. Healthy volunteers will be placed with a professional retrospective glucose monitoring device and will be tested for stimulation with arginine infusion. The device will be placed on the day of the test and will be removed after seven days of recording the glycemic data. During the entire recording period, parameters such as mean glucose, estimated glycosylated hemoglobin, peak glucose and nadir, blood sugar levels above the limit of 140 mg / dL, average glucose values at 60 and 120 minutes after meals, standard deviation and variability coefficient.
  Interventions: Diagnostic Test: Stimulation test with arginine infusion in order to verify the possible existence of damage to the beta cell function induced by COVID-19 infection
- Type 2 diabetes patients (Other): Patients with established Type 2 diabetes, not affects by COVID-19. Patients will be placed with a professional retrospective glucose monitoring device and will be tested for stimulation with arginine infusion. The device will be placed on the day of the test and will be removed after seven days of recording the glycemic data. During the entire recording period, parameters such as mean glucose, estimated glycosylated hemoglobin, peak glucose and nadir, blood sugar levels above the limit of 140 mg / dL, average glucose values at 60 and 120 minutes after meals, standard deviation and variability coefficient.
  Interventions: Diagnostic Test: Stimulation test with arginine infusion in order to verify the possible existence of damage to the beta cell function induced by COVID-19 infection

INTERVENTIONS:
Diagnostic Test: Stimulation test with arginine infusion in order to verify the possible existence of damage to the beta cell function induced by COVID-19 infection — All participants will be subjected to the collection of glycemic data through continuous professional retrospective monitoring of blood glucose for seven days, positioned on the day the test will be performed. During the entire recording period, parameters such as mean glucose, estimated glycosylated hemoglobin, peak glucose and nadir, blood sugar levels above the limit of 140 mg / dL, average glucose values at 60 and 120 minutes after meals, standard deviation and variability coefficient.
  The evaluation of insulin secretion will be evaluated by performing the stimulus test with arginine infusion according to validated protocols.
  Other Names: Positioning of the device for glycemic monitoring

SUMMARY:
In recent months, a new coronavirus, SARS-CoV-2, has been identified as the cause of a serious lung infection named COVID-19 by the World Health Organization. This virus has spread rapidly among the nations of the world and it is the cause of a pandemic and a global health emergency. There is still very little scientific evidence on the virus, however epidemiological data suggest that one of the most frequent comorbidities is diabetes, along with hypertension and heart disease. There is no scientific evidence on the possible effects of this infection on the function of the β cell and on glycemic control. Clinical evidence seems to suggest that COVID-19 infection mostly affects the respiratory system, and an acute worsening of glycemic compensation is not described as generally observed in bacterial pneumonia. However, previous work on acute respiratory syndromes (SARS) caused by similar coronaviruses, had described that the infection has multi-organ involvement related to the expression of the SARS coronavirus receptor, the angiotensin 2 converting enzyme, in different organs, especially at the level of endocrine pancreatic tissue. In the population of this previous work, glucose intolerance and fasting hyperglycaemia have been described and in 37 of 39 diabetic patients examined, a remission of diabetes was observed three years after the infection. It is possible that the coronaviruses responsible for SARS may enter the pancreatic islets using the angiotensin 2 converting enzyme receptor, expressed at the level of the endocrine pancreas, thus causing diabetes. Additionally, previous literature on coronavirus infections (SARS and MERS or Middle-East Respiratory Syndrome) suggested that diabetes could worsen the evolution of the disease. In particular, in case of Middle-East Respiratory Syndrome-CoV infection, diabetic mice had a more prolonged serious illness and a delay in recovery regardless of the viremic titer. This could probably be due to a dysregulation of the immune response, which results in more serious and prolonged lung disease.

There are currently no data on pancreatic beta cell function in patients with COVID-19.

DETAILED DESCRIPTION:
The project is monocentric, interventional, non-pharmacological, non-profit. Patients will be enrolled in hospital for confirmed COVID-19 infection (with reverse transcriptase-polymerase chain reaction on the airway swab) but with normal basal blood glucose and no previous history of diabetes or impaired fasting glucose or impaired glucose tolerance. Patients will be compared to a control group of healthy volunteers, not affected by COVID-19 and with no previous history of diabetes or impaired fasting glucose or impaired glucose tolerance. Patients will be also compared with a group of patients with type 2 diabetes but without COVID-19. Once the informed consent has been signed, the clinical parameters and biochemical parameters will be collected according to the time points provided by the protocol in positive COVID-19 patients, in healthy volunteers and in patients with type 2 diabetes.

COVID-19 positive patients and healthy controls as well as patients with type 2 diabetes, will undergo a stimulation test of β-cell function (evaluation of the secretive response of insulin to the stimulation test with arginine infusion) and the monitoring of glycemic values through a professional retrospective continuous glucose monitoring. For the test, an infusion solution containing 25% arginine hydrochloride will be used, arginine is an insulinogenic amino acid, useful to verify the possible existence of damage to the cellular beta function induced by COVID-19 infection, clinically observable with changes in insulin secretory response. Given the usefulness of the test, performed for diagnostic purposes, this protocol is identified as "non-pharmacological". The test is contraindicated only in patients with severe hepatic and renal insufficiency, in all other subjects the side effects are minimal and spontaneous resolution before the end of the test (flushing 33%, oral paraesthesia 46%, nausea 12%, dizziness 14%). For the stimulation test with arginine infusion, after the basal sampling at (0 minutes), an intravenous injection of arginine 5 grams will be practiced in 60 seconds followed by serial withdrawals at +2, +5, +10 and +30 minutes. The following analytes will be assayed on the basal sample: glycosylated hemoglobin, glycaemia, insulin, pro-insulin, C-peptide, glucagon, serum inflammatory cytokines (Il1β, IL-2, IL-6, IL-7, IL-10, TNF- α, IFN-γ, MIP-1β, MCP-1, GM-CSF, G-CSF Insulin, C-peptide and glucagon will be dosed on all points of the curve.

ELIGIBILITY:
Inclusion criteria for COVID-19 positive patients

* Male and female patients with COVID19 and normal basal blood sugar, unprecedented in diabetes or impaired fasting glucose or impaired glucose tolerance
* Age> 18 years and <80 years
* Availability to informed consent and corporate privacy

Inclusion criteria for healthy subjects

* Male and female patients not affected by COVID19, unprecedented in diabetes or impaired fasting glucose or impaired glucose tolerance
* Age> 18 years and <80 years
* Availability to informed consent and corporate privacy

Exclusion criteria for COVID-19 positive patients

* Age <18 years
* Previous history of diabetes or impaired fasting glucose or impaired glucose tolerance
* Severe liver failure
* Severe kidney failure

Exclusion criteria for healthy subjects

* Age <18 years
* Previous history of diabetes or impaired fasting glucose or impaired glucose tolerance
* Positivity to the nasopharyngeal swab for SARS-CoV-2
* Severe liver failure
* Severe kidney failure

Inclusion criteria for T2D patients

* Male and female patients not affected by COVID19 with a diagnosis of type 2 diabetes
* Age> 18 years and <80 years
* Availability to informed consent and corporate privacy

Exclusion criteria for T2D patients

* Age <18 years
* Positivity to the nasopharyngeal swab for SARS-CoV-2
* Severe liver failure
* Severe kidney failure

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2020-06-30 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Serum β - cellular function index insulin levels | all data were collected at Visit 1, 12 months
  Difference in insulin levels during and after COVID-19 infection and compared to patients in the control group
Serum β - cellular function index C-peptide levels | all data were collected at Visit 1, 12 months
  Difference in C-peptide levels during and after COVID-19 infection and compared to patients in the control group
Serum β - cellular function HOMA-β index | all data were collected at Visit 1, 12 months
  Difference in HOMA-β index during and after COVID-19 infection and compared to patients in the control group
Serum β - cellular function pro-insulin/insulin ratio | all data were collected at Visit 1, 12 months
  Difference in pro-insulin/insulin ratio during and after COVID-19 infection and compared to patients in the control group
Evaluation of the secretory response of insulin to the arginine stimulation test | all data were collected at Visit 1, 12 months
  Check for the existence of damage to the beta cell function induced by COVID-19 infection, clinically observable with changes in the secretory response of insulin
Percentage of patients with preserved β cells function | all data were collected at Visit 1, 12 months
  Evidence of impairment of β cell function in the serum of COVID-19 patients

SECONDARY OUTCOMES:
Glucose values | all data were collected at Visit 1, 12 months
  Changes in glucose values in COVID-19 patients and healthy volunteers
Values of continuous glucose monitoring | all data were collected at Visit 1 and after 7 days, 12 months
  Changes in the values of continuous glucose monitoring in both COVID-19 patients and healthy volunteers
Changes in the inflammatory marker interleukin 1-β | all data were collected at Visit 1, 12 months
  Comparison of interleukin 1-β levels in COVID-19 patients compared with healthy subjects
Changes in the inflammatory marker interleukin IL-2 | all data were collected at Visit 1, 12 months
  Comparison of interleukin IL-2 levels in COVID-19 patients compared with healthy subjects
Changes in the inflammatory marker interleukin IL-6 | all data were collected at Visit 1, 12 months
  Comparison of interleukin IL-6 levels in COVID-19 patients compared with healthy subjects
Changes in the inflammatory marker interleukin IL-7 | all data were collected at Visit 1, 12 months
  Comparison of interleukin IL-7 levels in COVID-19 patients compared with healthy subjects
Changes in the inflammatory marker interleukin IL-10 | all data were collected at Visit 1, 12 months
  Comparison of interleukin IL-10 levels in COVID-19 patients compared with healthy subjects
Changes in the inflammatory marker tumor necrosis factor-α | all data were collected at Visit 1, 12 months
  Comparison of interleukin tumor necrosis factor-α levels in COVID-19 patients compared with healthy subjects
Changes in the inflammatory marker interferon gamma | all data were collected at Visit 1, 12 months
  Comparison of interferon gamma levels in COVID-19 patients compared with healthy subjects
Changes in the inflammatory marker macrophage inflammatory protein-1β | all data were collected at Visit 1, 12 months
  Comparison of macrophage inflammatory protein-1β levels in COVID-19 patients compared with healthy subjects
Changes in the inflammatory marker monocyte chemoattractant protein-1 | all data were collected at Visit 1, 12 months
  Comparison of macrophage inflammatory monocyte chemoattractant protein-1 in COVID-19 patients compared with healthy subjects
Changes in the inflammatory marker granulocyte-macrophage colony-stimulating factor | all data were collected at Visit 1, 12 months
  Comparison of macrophage inflammatory granulocyte-macrophage colony-stimulating factor in COVID-19 patients compared with healthy subjects
Changes in the inflammatory marker granulocyte colony-stimulating factor | all data were collected at Visit 1, 12 months
  Comparison of macrophage inflammatory granulocyte colony-stimulating factor in COVID-19 patients compared with healthy subjects

CONTACTS AND LOCATIONS:
Locations (1):
- Sacco University Hospital, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Deng SQ, Peng HJ. Characteristics of and Public Health Responses to the Coronavirus Disease 2019 Outbreak in China. J Clin Med. 2020 Feb 20;9(2):575. doi: 10.3390/jcm9020575. PMID 32093211
- [Background] Kulcsar KA, Coleman CM, Beck SE, Frieman MB. Comorbid diabetes results in immune dysregulation and enhanced disease severity following MERS-CoV infection. JCI Insight. 2019 Oct 17;4(20):e131774. doi: 10.1172/jci.insight.131774. PMID 31550243
- [Background] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Background] Yang JK, Lin SS, Ji XJ, Guo LM. Binding of SARS coronavirus to its receptor damages islets and causes acute diabetes. Acta Diabetol. 2010 Sep;47(3):193-9. doi: 10.1007/s00592-009-0109-4. Epub 2009 Mar 31. PMID 19333547
- [Background] Shankar SS, Vella A, Raymond RH, Staten MA, Calle RA, Bergman RN, Cao C, Chen D, Cobelli C, Dalla Man C, Deeg M, Dong JQ, Lee DS, Polidori D, Robertson RP, Ruetten H, Stefanovski D, Vassileva MT, Weir GC, Fryburg DA; Foundation for the National Institutes of Health beta-Cell Project Team. Standardized Mixed-Meal Tolerance and Arginine Stimulation Tests Provide Reproducible and Complementary Measures of beta-Cell Function: Results From the Foundation for the National Institutes of Health Biomarkers Consortium Investigative Series. Diabetes Care. 2016 Sep;39(9):1602-13. doi: 10.2337/dc15-0931. Epub 2016 Jul 12. PMID 27407117
- [Background] Brandle M, Lehmann R, Maly FE, Schmid C, Spinas GA. Diminished insulin secretory response to glucose but normal insulin and glucagon secretory responses to arginine in a family with maternally inherited diabetes and deafness caused by mitochondrial tRNA(LEU(UUR)) gene mutation. Diabetes Care. 2001 Jul;24(7):1253-8. doi: 10.2337/diacare.24.7.1253. PMID 11423511
- [Derived] Bolla AM, Loretelli C, Montefusco L, Finzi G, Abdi R, Ben Nasr M, Lunati ME, Pastore I, Bonventre JV, Nebuloni M, Rusconi S, Santus P, Zuccotti G, Galli M, D'Addio F, Fiorina P. Inflammation and vascular dysfunction: The negative synergistic combination of diabetes and COVID-19. Diabetes Metab Res Rev. 2022 Oct;38(7):e3565. doi: 10.1002/dmrr.3565. Epub 2022 Jul 22. PMID 35830597
- [Derived] Ben Nasr M, D'Addio F, Montefusco L, Usuelli V, Loretelli C, Rossi A, Pastore I, Abdelsalam A, Maestroni A, Dell'Acqua M, Ippolito E, Assi E, Seelam AJ, Fiorina RM, Chebat E, Morpurgo P, Lunati ME, Bolla AM, Abdi R, Bonventre JV, Rusconi S, Riva A, Corradi D, Santus P, Clark P, Nebuloni M, Baldi G, Finzi G, Folli F, Zuccotti GV, Galli M, Herold KC, Fiorina P. Indirect and Direct Effects of SARS-CoV-2 on Human Pancreatic Islets. Diabetes. 2022 Jul 1;71(7):1579-1590. doi: 10.2337/db21-0926. PMID 35499468